CLINICAL TRIAL: NCT06563791
Title: Assessment of the Association Between Visceral Obesity and the Progression of Diabetic Nephropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourhan Mohamed Ehab Ahmed, Doctor, Assiut University
Other Study IDs: Visceral obesity and DN
Record Dates: First submitted 2024-08-06; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the association between visceral obesity and the progression of diabetic nephropathy

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a disorder of diverse aetiology characterised by hyperglycemia resulting from abnormalities of insulin action, insulin production, or both, and the global population with diabetes mellitus is expected to be around 439 million by 2030 . Diabetic nephropathy is the most prevalent microvascular consequence of DM. It develops in around 40% of DM patients.

Obesity, which has now reached pandemic ratios, is frequently accompanied by diabetes mellitus type 2 because they share common pathophysiological pathways . Abdominal obesity is found to be a negligent form of obesity with dangerous consequences. It has been identified as potentially hazardous factor for diabetic complications. Several abdominal obesity measures have been developed including the visceral adiposity index (VAI) , lipid accumulation product (LAP) , neck circumference (NC), waist-to-hip ratio (WHR) Lipid accumulation product (LAP) and visceral adiposity index (VAI) are new, non-imaging indicators of visceral adiposity measured using body mass index (BMI), waist circumference (WC), and serum lipid profile. It was predicted in some studies that LAP and VAI have a stronger association with poor renal outcomes than BMI and WC.

ELIGIBILITY:
Inclusion Criteria:

- 1. Diabetic patients either type 1 or type 2 diabetes aged > 18 years whether known to have diabetic nephropathy or not.

2. BMI is ≥ 25 kg/m2

Exclusion Criteria:

* 1. Patients age < 18 years. 2. BMI < 25 kg/m2 3. Nondiabetic patients 4. Patients with non-diabetic kidney disease. 5. Patients with AKI 6. Patients with CKD stage 5 either on dialysis or not.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients either type 1 or type 2 diabetes aged > 18 years whether known to have diabetic nephropathy or not with BMI is ≥ 25 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the association between visceral obesity and the progression of diabetic nephropathy | Baseline
  Assessment of visceral obesity new measures as (the visceral adiposity index (VAI) , lipid accumulation product (LAP) , neck circumference (NC), waist-to-hip ratio (WHR) ) as a risk factor for the progression of diabetic nephropathy and poor renal outcome.

REFERENCES:
- [Result] Thipsawat S. Early detection of diabetic nephropathy in patient with type 2 diabetes mellitus: A review of the literature. Diab Vasc Dis Res. 2021 Nov-Dec;18(6):14791641211058856. doi: 10.1177/14791641211058856. PMID 34791910
- [Result] Boutari C, DeMarsilis A, Mantzoros CS. Obesity and diabetes. Diabetes Res Clin Pract. 2023 Aug;202:110773. doi: 10.1016/j.diabres.2023.110773. Epub 2023 Jun 23. PMID 37356727
- [Result] Wan H, Wang Y, Xiang Q, Fang S, Chen Y, Chen C, Zhang W, Zhang H, Xia F, Wang N, Lu Y. Associations between abdominal obesity indices and diabetic complications: Chinese visceral adiposity index and neck circumference. Cardiovasc Diabetol. 2020 Jul 31;19(1):118. doi: 10.1186/s12933-020-01095-4. PMID 32736628
- [Result] Bullen AL, Katz R, Kumar U, Gutierrez OM, Sarnak MJ, Kramer HJ, Shlipak MG, Ix JH, Judd SE, Cushman M, Garimella PS. Lipid accumulation product, visceral adiposity index and risk of chronic kidney disease. BMC Nephrol. 2022 Dec 15;23(1):401. doi: 10.1186/s12882-022-03026-9. PMID 36522626